CLINICAL TRIAL: NCT02250339
Title: Phase 2: A Prospective Observational Study of Feasibility and Tentative Effectiveness of Multi-Systemic and Multicomponent Family-Based Intervention for Families of Children With Neuropsychiatric and/or Psychiatric Disorder(s).
Brief Title: A Prospective Observational Study of Family-based Interventions for Children With Neuropsychiatric and/or Psychiatric Disorders
Status: Completed | Type: Observational
Sponsor: Social Insurance Institution, Finland (Other)
Collaborators: Turku University Hospital (Other Government); University of Turku (Other)
Responsible Party: Sponsor
Other Study IDs: Perhe14; Kela (Other: The Social Insurance Institution of Finland)
Record Dates: First submitted 2014-09-18; First posted 2014-09-26 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2016-01

CONDITIONS: ADHD; Asperger Syndrome; Child Behavior Disorders
Keywords: Child Mental Health; Parenting; Family Issues
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Asperger Syndrome; Child Behavior Disorders | interventions — Family Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- LAKU family program: Time-limited (12 or 24 months) intervention program for children (aged 5-12) with neuropsychiatric/psychiatric disorder(s). LAKU family program (12 month program) includes 35 family-based meetings. Families are also given an opportunity to attend two separate family weekends. In addition to this, parent group format may include 10 meetings at maximum. A 24-month-program will include 15 additional family-based meetings.
  Interventions: Other: LAKU family program
- Etä-LAKU family program: Time-limited (18 or 24 months) intervention program for children (aged 5-12) with neuropsychiatric/psychiatric disorder(s). Etä-LAKU family program (18 months) includes 35 family-based meetings and two separate family weekends. A 24-month-program will include 10 additional family-based meetings.
  Interventions: Other: Etä-LAKU family program
- Family therapy: Time-limited (12 or 24 months) family therapeutic intervention for children (aged 5-12) with neuropsychiatric/psychiatric disorder(s). Family therapy intervention includes 15 (1-year program) or 30 (2-year program) family meetings.
  Interventions: Other: Family therapy

INTERVENTIONS:
Other: LAKU family program — Multi-systemic and multicomponent family-based intervention program
  Groups: LAKU family program
Other: Etä-LAKU family program — Ecosystem-based intervention for families living in rural parts of Finland
  Groups: Etä-LAKU family program
Other: Family therapy — Treatment as usual (TAU)
  Groups: Family therapy

SUMMARY:
The purpose of this study is to examine the feasibility and the effects of family-based interventions for children (aged 5-12) with neuropsychiatric and psychiatric disorders in Finnish health care settings.

DETAILED DESCRIPTION:
1. Introduction

   The role of the Social Insurance Institution of Finland (Kela) is to complement publicly funded Finnish health care delivery system. In 2003, the Finnish Ministry of Social Affairs and Health further defined that Kela fund mental health services for children under 16 years old should incorporate family oriented psychological counselling and multicomponent rehabilitation. The purpose of the present prospective observational study is to examine the feasibility and tentative effectiveness of a multi-systemic and multicomponent family interventions for 5-12 year-old children with neuropsychiatric symptoms. The present study design is defined by the following key characteristics: (a) it comprises the comparison of three clinically relevant interventions based on family therapeutic activities; (b) it involves a diverse population of participants from heterogeneous practice settings; and (c) intervention outcomes are defined relatively broadly. All study participants will be recruited in Finland. The research is also conducted in Finland by the Finnish research consortium. The research project is funded by the Health department of the Social Insurance Institution of Finland.
2. Effectiveness of family-systemic interventions for children with mental health problems

   Empirical evidence supports the effectiveness of family-systemic and family-based interventions for children who may suffer from, for example, socio-emotional and developmental problems that relate to neuropsychiatric disorders such as ADHD and Autism Spectrum Disorder. Family-systemic interventions may, firstly, refer to a more traditional and distinct method of psychotherapy (i.e. family therapy) provided by a licensed therapist. Secondly, the family systemic and therapeutic approach has further influenced the development and implementation of specific licensed family-focused and empirically supported treatment program protocols (e.g. MST and MDFT). Thirdly, there are also specific behavioral and cognitive-behavioral parent training protocols available (e.g. PMTO and Triple P), which are considered a form of family-based approach. However, the rationale in parent training protocols stems more solely from social learning theory and interventions are typically delivered in a parent group format. It could be further argued that family-focused treatment protocols and parent training programs reflect the emergence of a so-called third-generation family therapeutic perspective by enhancing the need to establish evidence-based interventions through randomized controlled clinical trials. In addition to discussions above, family therapy is the most popular therapy approach among licensed psychotherapists working in the health care system in Finland. However, there is very little research on the effects of family-systemic interventions on the well-being of children with mental health problems and their families in Finnish health care settings.
3. Description of the interventions

   The multi-systemic and multicomponent family intervention for 5-12 year-old children with neuropsychiatric symptoms is based on the intervention program developed by the Health department of the Social Insurance Institution of Finland. In order to incorporate the best current practices and delivery formats, an independent expert panel of child psychiatry specialists from the Finnish University Hospitals was recruited in intervention development. Intervention feasibility and acceptability were further assessed by piloting work. At the present project, time-limited services (12 to 24 months) are provided in two different arms (i.e. separate intervention programs) referred to as LAKU and Etä-LAKU family intervention programs. Aims of the family intervention are to help children to strengthen their socio-emotional skills at home and in everyday life settings, help children and families to cope with their experiences, and strengthen interpersonal interaction among family members to overcome possibly difficult life situations, thoughts and emotions.

   The family therapeutic approach is the key intervention component. Family sessions are provided by a licensed family therapist and a co-worker who is also an experienced mental health care professional. Multi-systemic approach addresses the importance of individualized needs of children and families. This includes the work with other important social systems (e.g. child daycare and school). The multi-systemic approach also includes both visiting and monitoring the child in his/hers social environment as well as collaborative meetings together with the family and the child's significant others from daycare and school. The collaborative stance further requires that family workers attach assigned family consultants from the health care delivery system as part of the therapeutic system too. The multicomponent approach, for its part, is designed to provide different delivery formats for the families involved such as group meetings for parents. Other important delivery formats include one-to-one sessions with the child. The families are also given an opportunity to attend family weekends where they can meet other families who share similar life situations.

   LAKU and Etä-LAKU family intervention programs have some pertinent differences. The prior intervention program is provided in an 'urban' context and therapeutic sessions may take place flexibly both at a clinic and in the family's home. Etä-LAKU, however, is strictly an ecosystem-based family intervention program. It is tailored for families who live in rural parts of Finland with very limited health services available. The Etä-LAKU family intervention program does not include the delivery of parent group sessions either. The LAKU family program involves service providers and child mental health clinics in the Finnish towns of Helsinki, Kotka, Tampere and Oulu as well as their environs. The Etä-LAKU intervention program is provided in Lapland and Kainuu/Ylä-Savo environs.
4. Prospective observational clinical study

The centerpiece of the project will be a prospective observational study of 5-12 year-old children and their parents who attend family-systemic interventions in different practical settings. The observational study is further based on multisource (i.e. child, parent and teacher report) assessment design. The study has been approved by the Research Ethics Committee of the Hospital District of Southwest Finland and the Research Ethics Committee of the Kela research department. Study approval from the Hospital District of Southwest Finland is in process.

The control group consists of children and families attending family therapy. Time-limited family therapy (12 to 24 months) is provided via the Hospital District of Southwest Finland/Turku University Hospital's Child Psychiatry clinic (TYKS) and takes place in the town of Turku environs. All data will be collected in Finland and stored at the Research department of the Social Insurance Institution of Finland, located in Helsinki. Study measures will be administered in Finnish only.

The study design does not include randomization. However, it provides an opportunity to compare possible changes in child and parent well-being within and between three different and clinically relevant family intervention programs. Beyond this, key outcome variables are determined by giving the possibility to scrutinize intervention effectiveness more closely. The study design enables comparing the results from primary and secondary outcomes to those from nationally representative school- and population-based surveys conducted in Finland.

ELIGIBILITY:
Inclusion Criteria:

* Child is 5-12 year-old at time of recruitment
* Child meets screening criteria for neuropsychiatric disorder (i.e. ADHD & Asperger Syndrome)
* Child may also meet screening criteria for co-existing condition such as Behavior Disorder
* Family situation is assessed by the health care professional (child psychiatrist) and an intensive family-based intervention is further recommended

Exclusion Criteria:

* Child's psychiatric condition requires acute inpatient care
* Child's parent's alcohol and/or substance abuse requires acute treatment
* The progress is going on to correct the conditions that may lead to the child's placement in out-of-home care

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The LAKU family program service is provided in Helsinki, Kotka, Tampere and Oulu environs. The Etä-LAKU intervention program is provided in Lapland and Kainuu/Ylä-Savo environs. Families are admitted to the programs by the child mental health clinics in the respective localities. The control group (treatment as usual) consists of children and families attending the family therapy fund by the Hospital District of Southwest Finland/Turku University Hospital's Child Psychiatry clinic (TYKS) and takes place in the Hospital District of Southwest Finland environs. Potential participants (i.e. the families admitted to the family-based intervention) will receive both oral and written information about the study and an invitation to volunteer. Both parents (when applicable) and child are advised to participate independently. Power analysis is utilized to ensure minimum necessary number of study participants. Anticipated sample sizes are: n=125 (LAKU), n=72 (Etä-LAKU), and n=33 (TAU group).
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Child's Health Related Quality of Life questionnaire (HRQOL) - (KINDL-R) | Participants will be followed to measure change from baseline to an expected average of 12-18 months & 24 months (when applicable) + 6 months post-intervention follow-up
  KINDL-R is a generic instrument, which involves both child and parent reports.
Multisource Assessment of Children's Socioemotional Competence Scale (MASCS) | Participants will be followed to measure change from baseline to an expected average of 12-18 months & 24 months (when applicable) + 6 months post-intervention follow-up
  The MASCS is developed on the of The School Social Behavior Scales (SSBS), and it measures child's prosocial and antisocial behaviour. Multisource assessment includes child, parent and teacher reports.
Parenting Self-Efficacy (PSE) | Participants will be followed to measure change from baseline to an expected average of 12-18 months & 24 months (when applicable) + 6 months post-intervention follow-up
  The PSE is a Finnish modification version of the Self-Efficacy for Parenting Tasks Index (SEPTI).

SECONDARY OUTCOMES:
Finnish version of the Peer Network and Dyadic Loneliness Scale (PNDL) | Participants will be followed to measure change from baseline to an expected average of 12-18 months & 24 months (when applicable) + 6 months post-intervention follow-up
  PNDL measures lack of involvement in a social network and the absence of close dyadic friendships. Child report only.
Mental Health Inventory (MHI-5) | Participants will be followed to measure change from baseline to an expected average of 12-18 months & 24 months (when applicable) + 6 months post-intervention follow-up
  To measure for Parent's Psychological Stress

OTHER OUTCOMES:
Parenting and Family Life Related Stress Measures | Participants will be followed to measure change from baseline to an expected average of 12-18 months & 24 months (when applicable)+ 6 months post-intervention follow-up
  Participants will be followed to measure psychological stress that stems from family related issues. Items are derived from Finnish family surveys conducted by the National Institute for Health and Welfare.
Satisfaction measures | Satisfaction will be measured at the end of an expected program average of 12-18 months & 24 months (when applicable)
  To measure intervention acceptability and feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Miika Vuori, Ph.D., Principal Investigator — Research Department, Social Insurance Institution of Finland
Locations (1):
- Social Insurance Institution, Helsinki, Finland

REFERENCES:
- [Background] Littell JH, Popa M, Forsythe B. Multisystemic Therapy for social, emotional, and behavioral problems in youth aged 10-17. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD004797. doi: 10.1002/14651858.CD004797.pub3. PMID 16034952
- [Background] Barlow J, Smailagic N, Huband N, Roloff V, Bennett C. Group-based parent training programmes for improving parental psychosocial health. Cochrane Database Syst Rev. 2014 May 17;2014(5):CD002020. doi: 10.1002/14651858.CD002020.pub4. PMID 24838729
- [Background] Gross DA, Belcher HM, Ofonedu ME, Breitenstein S, Frick KD, Chakra B. Study protocol for a comparative effectiveness trial of two parent training programs in a fee-for-service mental health clinic: can we improve mental health services to low-income families? Trials. 2014 Mar 1;15:70. doi: 10.1186/1745-6215-15-70. PMID 24581245
- [Background] Lee PC, Niew WI, Yang HJ, Chen VC, Lin KC. A meta-analysis of behavioral parent training for children with attention deficit hyperactivity disorder. Res Dev Disabil. 2012 Nov-Dec;33(6):2040-9. doi: 10.1016/j.ridd.2012.05.011. Epub 2012 Jun 29. PMID 22750360
- [Background] Charach A, Carson P, Fox S, Ali MU, Beckett J, Lim CG. Interventions for preschool children at high risk for ADHD: a comparative effectiveness review. Pediatrics. 2013 May;131(5):e1584-604. doi: 10.1542/peds.2012-0974. Epub 2013 Apr 1. PMID 23545375
- [Background] Zwi M, Jones H, Thorgaard C, York A, Dennis JA. Parent training interventions for Attention Deficit Hyperactivity Disorder (ADHD) in children aged 5 to 18 years. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD003018. doi: 10.1002/14651858.CD003018.pub3. PMID 22161373
- [Background] Reyno SM, McGrath PJ. Predictors of parent training efficacy for child externalizing behavior problems--a meta-analytic review. J Child Psychol Psychiatry. 2006 Jan;47(1):99-111. doi: 10.1111/j.1469-7610.2005.01544.x. PMID 16405646
- [Background] Lundahl B, Risser HJ, Lovejoy MC. A meta-analysis of parent training: moderators and follow-up effects. Clin Psychol Rev. 2006 Jan;26(1):86-104. doi: 10.1016/j.cpr.2005.07.004. Epub 2005 Nov 8. PMID 16280191
- [Background] Shepperd S, Doll H, Gowers S, James A, Fazel M, Fitzpatrick R, Pollock J. Alternatives to inpatient mental health care for children and young people. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD006410. doi: 10.1002/14651858.CD006410.pub2. PMID 19370634
- [Background] Carr, A. (2014), The evidence base for family therapy and systemic interventions for child-focused problems. Journal of Family Therapy, 36: 107-157. doi: 10.1111/1467-6427.12032
- [Background] Dunst CJ, Trivette CM, Hamby DW. Meta-analysis of family-centered helpgiving practices research. Ment Retard Dev Disabil Res Rev. 2007;13(4):370-8. doi: 10.1002/mrdd.20176. PMID 17979208
- [Background] Robin AL. Family therapy for adolescents with ADHD. Child Adolesc Psychiatr Clin N Am. 2014 Oct;23(4):747-56. doi: 10.1016/j.chc.2014.06.001. Epub 2014 Aug 8. PMID 25220084
- [Background] Kolko DJ, Campo J, Kilbourne AM, Hart J, Sakolsky D, Wisniewski S. Collaborative care outcomes for pediatric behavioral health problems: a cluster randomized trial. Pediatrics. 2014 Apr;133(4):e981-92. doi: 10.1542/peds.2013-2516. Epub 2014 Mar 24. PMID 24664093
- [Background] Karst JS, Van Hecke AV. Parent and family impact of autism spectrum disorders: a review and proposed model for intervention evaluation. Clin Child Fam Psychol Rev. 2012 Sep;15(3):247-77. doi: 10.1007/s10567-012-0119-6. PMID 22869324
- [Background] Matson JL, Mahan S, LoVullo SV. Parent training: a review of methods for children with developmental disabilities. Res Dev Disabil. 2009 Sep-Oct;30(5):961-8. doi: 10.1016/j.ridd.2009.01.009. Epub 2009 Feb 25. PMID 19246176
- [Background] Patterson SY, Smith V, Mirenda P. A systematic review of training programs for parents of children with autism spectrum disorders: single subject contributions. Autism. 2012 Sep;16(5):498-522. doi: 10.1177/1362361311413398. Epub 2012 Jan 16. PMID 22250194
- [Background] Danckaerts M, Sonuga-Barke EJ, Banaschewski T, Buitelaar J, Dopfner M, Hollis C, Santosh P, Rothenberger A, Sergeant J, Steinhausen HC, Taylor E, Zuddas A, Coghill D. The quality of life of children with attention deficit/hyperactivity disorder: a systematic review. Eur Child Adolesc Psychiatry. 2010 Feb;19(2):83-105. doi: 10.1007/s00787-009-0046-3. Epub 2009 Jul 26. PMID 19633992
- [Background] Cappe E, Wolff M, Bobet R, Adrien JL. Quality of life: a key variable to consider in the evaluation of adjustment in parents of children with autism spectrum disorders and in the development of relevant support and assistance programmes. Qual Life Res. 2011 Oct;20(8):1279-94. doi: 10.1007/s11136-011-9861-3. Epub 2011 Feb 12. PMID 21312064
- [Background] Rambo A, West C, Schooley AL, Boyd TV. (Eds). Family therapy review: Contrasting contemporary models. New York: Taylor and Francis. 2013.
- [Background] Rasheed JM, Rasheed MN, Marley JA. Family Therapy: Models and Techniques. London: SAGE.